CLINICAL TRIAL: NCT00006150
Title: Natural History, Management, and Genetics of the Hyperimmunoglobulin E Recurrent Infection Syndrome (HIES)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000159; 00-I-0159
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-07-08

CONDITIONS: Infections; Pneumonia; Immune System Diseases; STAT3 Transcription Factor; Job Syndrome
Keywords: DOCK8 Deficiency; PGM3 Deficiency; STAT3 Mutation; Job's Syndrome; Immunodeficiency; Natural History; Hyperimmunologobulin E Syndrome; HIE Syndrome
MeSH Terms: conditions — Infections; Pneumonia; Immune System Diseases; Job Syndrome; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected adults and children: Confirmed or suspected history of a Hyper IgE syndrome
- Relatives: Family members of subjects with confirmed or suspected history of a Hyper IgE syndrome

SUMMARY:
The Hyper IgE Syndromes (HIES) are primary immunodeficiencies resulting in eczema and recurrent skin and lung infections. Autosomal dominant Hyper IgE syndrome (AD-HIIES; Job's syndrome) is caused by STAT3 mutations, and is a multi-system disorder with skeletal, vascular, and connective tissue manifestations. Understanding how STAT3 mutations cause these diverse clinical manifestations is critical to our complete understanding of bone metabolism, bronchiectasis, dental maturation, and atherosclerosis. Bi-allelic mutations in DOCK8 cause a combined immunodeficiency previously described as autosomal-recessive Hyper IgE syndrome. These individuals suffer from extensive viral infections as well as have a high incidence of malignancy and mortality. The pathogenesis of this disease and long-term natural history is being investigated. Therefore, we seek to enroll patients and families with a confirmed or suspected diagnosis of HIES syndrome for extensive phenotypic and genotypic study as well as disease management. Patients will be carefully examined by a multidisciplinary team and followed longitudinally. Through these studies we hope to better characterize the clinical presentation of STAT3-mutated HIES, DOCK8 deficiency and other causes of the hyper IgE phenotype, and to be able to identify further genetic etiologies, as well as understand the pathogenesis of HIES. We seek to enroll 300 patients and 300 relatives....

DETAILED DESCRIPTION:
The Hyper IgE Syndromes (HIES) are primary immunodeficiencies resulting in eczema and recurrent skin and lung infections. Autosomal dominant Hyper IgE syndrome (AD-HIES; Job's syndrome) is caused by STAT3 mutations, and is a multi-system disorder with skeletal, vascular, and connective tissue manifestations. Understanding how STAT3 mutations cause these diverse clinical manifestations is critical to our complete understanding of bone metabolism, bronchiectasis, dental maturation, and atherosclerosis. Bi-allelic mutations in DOCK8 cause a combined immunodeficiency previously described as autosomal-recessive Hyper IgE syndrome. These individuals suffer from extensive viral infections as well as have a high incidence of malignancy and mortality. The pathogenesis of this disease and long-term natural history is being investigated. Therefore, we seek to enroll patients and families with a confirmed or suspected diagnosis of HIES syndrome for extensive phenotypic and genotypic study as well as disease management. Patients will be carefully examined by a multidisciplinary team and followed longitudinally. Through these studies we hope to better characterize the clinical presentation of STAT3-mutated HIES, DOCK8 deficiency and other causes of the hyper IgE phenotype, and to be able to identify further genetic etiologies, as well as understand the pathogenesis of HIES. We seek to enroll 300 patients and 300 relatives.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients may be included in this study who:

* Were referred to the NIH with a diagnosis or a suspicion of Hyper IgE syndrome.
* Are patients referred for other immune syndromes that demonstrate some of the characteristics of HIES.
* Are male or female, aged

Aged

* >=1 month for affected subjects
* Aged >=2 years for unaffected subjects

  * For unaffected subjects, are able to understand and have the willingness to sign a written informed consent document.

Unaffected biological relatives of HIES patients are also eligible to enroll in a separate relative cohort.

EXCLUSION CRITERIA:

Coronary CTA will not be performed on any patient younger than 30 years or with contraindication to IV contrast media. This includes patients with 1) creatinine value of >1.3 mg/dL, 2) history of multiple myeloma, 3) Use of metformin-containing products less than 24 hours prior to contrast media, and 4) history of significant allergic reaction to CT contrast agents despite the use of premedication.

Subjects with a medical, psychiatric, or social condition which, in the opinion of the investigator, would place undue burden on the subject, NIH resources, or increase risk of participation, may be excluded.

Ages: 1 Month to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2000-08-10 (Actual)

PRIMARY OUTCOMES:
To clinically phenotype AD-HIES, DOCK8 deficiency, PGM3 deficiency and other related hyper IgE syndromes | end of study
  established clinical phenotype of AD-HIES, DOCK8 deficiency, PGM3 deficiency and other related hyper IgE syndromes
To assess quality of life on the basis of clinical and immunologic evaluations | end of study
  quality of life assessments based on clinical and immunologic evaluations
To understand the pathogenesis of the immunologic defect in hyper IgE syndromes as well as the diverse clinical features such as wound healing abnormalities | end of study
  understanding of the pathogenesis of the immunologic defect in hyper IgE syndromes as well as the diverse clinical features such as wound healing abnormalities
To identify, characterize, and treat complications of the hyper IgE syndromes as they arise | end of study
  identification, characterization, and treatment of complications of the hyper IgE syndromes
To identify novel genetic defects leading to hyper IgE syndromes. | end of study
  identified novel genetic defects leading to hyper IgE syndromes.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra F Freeman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this study for future research as follows:@@@@@@@@@@@@Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC)@@@@@@@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements@@@@@@@@@@@@Data will be shared through: @@@@@@@@@@@@BTRIS (automatic for activities in the NIH CC)@@@@@@@@@@@@Approved outside collaborators under appropriate individual agreements@@@@@@@@@@@@Publication and/or public presentations.@@@@@@@@@@@@Data might be shared before publication.
Supporting Information: Study Protocol, ICF
Time Frame: IPD is available in real time in BTRIS.
Access Criteria: Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC) are available indefinitely.@@@@@@@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements

REFERENCES:
- [Background] Sowerwine KJ, Holland SM, Freeman AF. Hyper-IgE syndrome update. Ann N Y Acad Sci. 2012 Feb;1250:25-32. doi: 10.1111/j.1749-6632.2011.06387.x. Epub 2012 Jan 23. PMID 22268731
- [Background] Freeman AF, Holland SM. Clinical manifestations of hyper IgE syndromes. Dis Markers. 2010;29(3-4):123-30. doi: 10.3233/DMA-2010-0734. PMID 21178271
- [Background] Freeman AF, Avila EM, Shaw PA, Davis J, Hsu AP, Welch P, Matta JR, Hadigan C, Pettigrew RI, Holland SM, Gharib AM. Coronary artery abnormalities in Hyper-IgE syndrome. J Clin Immunol. 2011 Jun;31(3):338-45. doi: 10.1007/s10875-011-9515-9. Epub 2011 Apr 15. PMID 21494893
- [Background] Freeman AF, Collura-Burke CJ, Patronas NJ, Ilcus LS, Darnell D, Davis J, Puck JM, Holland SM. Brain abnormalities in patients with hyperimmunoglobulin E syndrome. Pediatrics. 2007 May;119(5):e1121-5. doi: 10.1542/peds.2006-2649. Epub 2007 Apr 16. PMID 17438082
- [Background] Grimbacher B, Holland SM, Gallin JI, Greenberg F, Hill SC, Malech HL, Miller JA, O'Connell AC, Puck JM. Hyper-IgE syndrome with recurrent infections--an autosomal dominant multisystem disorder. N Engl J Med. 1999 Mar 4;340(9):692-702. doi: 10.1056/NEJM199903043400904. PMID 10053178
- [Background] Holland SM, DeLeo FR, Elloumi HZ, Hsu AP, Uzel G, Brodsky N, Freeman AF, Demidowich A, Davis J, Turner ML, Anderson VL, Darnell DN, Welch PA, Kuhns DB, Frucht DM, Malech HL, Gallin JI, Kobayashi SD, Whitney AR, Voyich JM, Musser JM, Woellner C, Schaffer AA, Puck JM, Grimbacher B. STAT3 mutations in the hyper-IgE syndrome. N Engl J Med. 2007 Oct 18;357(16):1608-19. doi: 10.1056/NEJMoa073687. Epub 2007 Sep 19. PMID 17881745
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-I-0159.html